CLINICAL TRIAL: NCT05897333
Title: Turkish Isolated Coronary Ectasia Prospective Cohort Study: the T-ICE Registry
Brief Title: Turkish Isolated Coronary Ectasia Registry: The T-ICE Registry
Acronym: T-ICE
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Adnan Abacı, MD, Prof. Dr., Gazi University
Other Study IDs: 03063806
Record Dates: First submitted 2023-02-22; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated coronary ectasia: Includes the patients with isolated coronary artery ectasia without coronary stenosis.
- Coronary artery disease: Includes the patients with ≥50% stenosis in a vessel ≥2 mm in diameter.

SUMMARY:
The T-ICE study is a prospective, observational study aiming to have information about the treatment and long-term prognosis of patients with isolated coronary artery ectasia.

DETAILED DESCRIPTION:
Coronary artery ectasia is a localized or diffuse enlargement of the coronary artery lumen ≥1.5-2 times relative to the normal segment. It is often associated with coronary artery stenosis. Some patients have coronary artery ectasia without stenosis. This condition is called as isolated coronary artery ectasia. There is data other than retrospective studies with a small number of cases on the clinical significance, prognosis and treatment of isolated coronary ectasia in patients with or without acute coronary syndrome. Therefore, the treatment of patients with isolated coronary ectasia is not evidence-based and is based on the clinical judgment of physicians. The aim of this prospective observational study is to evaluate the treatment and prognosis of the isolated coronary artery ectasia. The second aim is to compare the prognosis of isolated coronary ectasia with the coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Isolated coronary artery ectasia (without ≥20% stenosis in any coronary artery ≥2 mm in diameter).
* All patients with isolated coronary ectasia with or without acute coronary syndrome will be included.
* Patients aged ≥18 years.
* Patients with discrete coronary artery aneurysm will be included.

Exclusion Criteria:

* Life expectancy <24 months
* Patients with ≥20% stenosis in a vessel ≥2 mm in diameter.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with "isolated" coronary ectasia in at least one coronary artery in their first coronary angiography performed for any reason will be included in the study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2032-03-15 (Estimated); Study Completion 2032-03-15 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events | Five years
  A composite endpoint of death, myocardial infarction, unstable angina, stroke, and coronary revascularization.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | Five years
  A composite endpoint of cardiovascular death, myocardial infarction, unstable angina, and coronary revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Abaci, Principal Investigator — Gazi University, School of Medicine, Department of Cardiology
Locations (1):
- Gazi University, School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manginas A, Cokkinos DV. Coronary artery ectasias: imaging, functional assessment and clinical implications. Eur Heart J. 2006 May;27(9):1026-31. doi: 10.1093/eurheartj/ehi725. Epub 2006 Jan 16. PMID 16415301
- [Background] Baman TS, Cole JH, Devireddy CM, Sperling LS. Risk factors and outcomes in patients with coronary artery aneurysms. Am J Cardiol. 2004 Jun 15;93(12):1549-51. doi: 10.1016/j.amjcard.2004.03.011. PMID 15194034
- [Background] Malviya A, Jha PK, Mishra A. Isolated coronary artery ectasia: Clinical, angiographic, and follow up characteristics. Indian Heart J. 2017 Sep-Oct;69(5):619-623. doi: 10.1016/j.ihj.2016.12.017. Epub 2017 Jan 22. PMID 29054186
- [Background] Erden I, Erden EC, Ozhan H, Karabulut A, Ordu S, Yazici M. Outcome of primary percutaneous intervention in patients with infarct-related coronary artery ectasia. Angiology. 2010 Aug;61(6):574-9. doi: 10.1177/0003319709361197. Epub 2010 Apr 14. PMID 20395236
- [Background] Vasu N, Narayanan S, Ajit MS. Clinical outcome of various management strategies in coronary artery ectasia. Indian Heart J. 2017 May-Jun;69(3):319-321. doi: 10.1016/j.ihj.2017.04.013. Epub 2017 May 4. No abstract available. PMID 28648421
- [Background] Boles U, Zhao Y, Rakhit R, Shiu MF, Papachristidis A, David S, Koganti S, Gilbert T, Henein MY. Patterns of coronary artery ectasia and short-term outcome in acute myocardial infarction. Scand Cardiovasc J. 2014 Jun;48(3):161-6. doi: 10.3109/14017431.2014.902495. Epub 2014 Apr 10. PMID 24673382
- [Background] Willner NA, Ehrenberg S, Musallam A, Roguin A. Coronary artery ectasia: prevalence, angiographic characteristics and clinical outcome. Open Heart. 2020 Apr;7(1):e001096. doi: 10.1136/openhrt-2019-001096. PMID 32515749